CLINICAL TRIAL: NCT03336996
Title: Assessement the Reconstruction of Motor Circuits in Nerve Fiber Injuries After the Treatment of Umbilical Cord Mesenchymal Stem Cells With Blood Oxygen Level-dependent Drived Diffusion Tensor Imaging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Xhechun4
Record Dates: First submitted 2017-10-26; First posted 2017-11-08 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-10

CONDITIONS: Characterize and Evaluate Functional After Transplantation; Determine the Therapeutic Efficiency; Correlate the Imaging Results
Keywords: Motor nerve injury; umbilical cord interstitial stem cell; bold-DTI; reconstruction of motor circuits
MeSH Terms: interventions — Stem Cell Transplantation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- evaluation (Experimental): To characterize and evaluate functional and anatomical changes of nerve fiber injuries after umbilical cord mesenchymal stem cells transplantation with BOLD drived-DTI
  Interventions: Procedure: BOLD-fMRI drived DTI scanning
- BOLD-fMRI and DTI (Experimental): To determine the therapeutic efficiency of umbilical cord mesenchymal stem cells and also the utility of the integration of BOLD-fMRI and DTI.
  Interventions: Biological: stem cell transplantation
- correlate the imaging results (Experimental): To correlate the imaging results with the electrophysiology outcomes
  Interventions: Procedure: BOLD-fMRI drived DTI scanning

INTERVENTIONS:
Biological: stem cell transplantation — the motor nerve fiber damaged patient receive a treatment course stem cell transplantation after the hematoma removal.
  Arms: BOLD-fMRI and DTI
Procedure: BOLD-fMRI drived DTI scanning — All patients should be receive cranial BOLD-fMRI drived DTI scanning scanning separately before the transplant and after the transplant 0, 1, 3, 6 and 12 months.
  Arms: correlate the imaging results; evaluation

SUMMARY:
Nowadays, the stem cell therapy is a promising method in treatment of the traumatic nerve fiber injuries. And the clinical use of umbilical cord mesenchymal stem cells has been approved by FDA. However, the results are inconsistent from both human study and animal research, it often difficult to visualize the reconstruction of the motor circuits. A separate application of DTI could not precisely reveal white matter integrity. Combining blood oxygen level-dependent(BOLD)-functional magnetic resonance imaging(fMRI) with diffusion tensor-based tractography (DTT), to detect neural activities in the brain involved in the motor function restore and then using the two seeds method to reconstruct the nerve fibers between these connecting regions. The main aim of this study: i. To characterize and evaluate functional and anatomical changes of nerve fiber injuries after umbilical cord mesenchymal stem cells transplantation with BOLD drived-diffusion tensor imaging(DTI). ii. To determine the therapeutic efficiency of umbilical cord mesenchymal stem cells and also the utility of the integration of BOLD-fMRI and DTI. iii. To correlate the imaging results with the electrophysiology outcomes.

DETAILED DESCRIPTION:
The stem cell therapy is a promising method in treatment of the traumatic nerve fiber injuries. And the clinical use of umbilical cord mesenchymal stem cells has been approved by FDA. However, the results are inconsistent from both human study and animal research, it often difficult to visualize the reconstruction of the motor circuits. A separate application of DTI could not precisely reveal white matter integrity. Combining BOLD-fMRI with diffusion tensor-based tractography (DTT), to detect neural activities in the brain involved in the motor function restore and then using the two seeds method to reconstruct the nerve fibers between these connecting regions. The main aim of this study: i. To characterize and evaluate functional and anatomical changes of nerve fiber injuries after umbilical cord mesenchymal stem cells transplantation with BOLD drived-DTI. ii. To determine the therapeutic efficiency of umbilical cord mesenchymal stem cells and also the utility of the integration of BOLD-fMRI and DTI. iii. To correlate the imaging results with the electrophysiology outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. All tested patients must be Sobriety and coordination the examination.
2. All tested patients with motor nerve fiber damaged must tally with the diagnosis standard which after the head CT, fMRI confirmation and obvious clinical symptoms.
3. Patient's age and gender: 20-65years，the gender is not limit;
4. All patient's must has one side neurological deficits.
5. The patient must receive surgery and stem cell transplantation.

Exclusion Criteria:

1. Progressive dysfunction;
2. Other internal organs strict illness sickness, like serious heart disease, diabetes, liver, kidney vigorous sickness and so on;
3. The patient with tumor in every system on there body;
4. Having the primary or the sequential epilepsy medical history, within one year had the epileptic paroxysm;
5. Can not accept MRI inspection, for some metal implant in there body(such as inner support in heart or brain blood vessel)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
BOLD-fMRI drived DTI scanning | After the transplant 6 months
  All patients should be receive cranial BOLD-fMRI drived DTI scanning scanning after the transplant 6 months, and the result tells us that there is obvious reconstruction of motor circuits in nerve fiber on the damaged region;

SECONDARY OUTCOMES:
FIM | after the transplant 6 months
  All patients should receive the function independence evaluation (FIM) after the transplant 6 months , and the grading has the distinct improvement;
NIHSS | after the transplant 6 months
  All patients should receive the American State-run Health Research institute apoplexy meter (NIHSS) evaluation after the transplant 6 months , and the grading has the distinct improvement;
Motor evoked potential | after the transplant 6 months
  All patients should be receive motor evoked potential after the transplant 6 months, and the function of movement and sensation get obvious improvement;

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: No